CLINICAL TRIAL: NCT05421975
Title: EASY MRI: Evaluating Airway Sarcoidosis Pathology With MRI
Brief Title: Evaluating Airway Sarcoidosis Pathology With MRI
Acronym: EASY MRI
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH21669
Record Dates: First submitted 2022-06-06; First posted 2022-06-16 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sarcoidosis is a condition where inflamed cells clump together to form granulomas, which can lead to inflammation or scarring. It can affect any organ of the body, but most commonly affects the lungs. Symptoms can be highly variable, and some patients have no symptoms where as others may develop fatigue or breathlessness. The causes of sarcoidosis are poorly understood. It commonly affects adults in their 30's or 40's.

Some patients present with symptoms suggestive of involvement in the airways, such as cough. Inhalers containing steroid are commonly used, but there is a poor understanding of which patients may benefit. Part of the problem is the lack of a sensitive way of measuring these effects and knowledge of how sarcoidosis affects the airways physiologically.

The investigators would like to know more about the disease process of sarcoidosis, particularly where it involves the airways. This study will use a number of techniques in order to better understand to disease process.

In order to assess whether sarcoidosis produces changes in airway ventilation (and whether these changes are stable or change over a short time period). This pilot study aims to recruit 6 patients who will have magnetic resonance imaging (MRI) with inhaled xenon gas. During this technique, xenon and nitrogen mixture is inhaled and during a subsequent breath-hold, images of the lungs are taken. This creates a detailed view of the lung airway tree, to explore how the disease affects the airways and deeper lung tissue.

This technique will be used alongside lung function tests, commonly performed in the laboratory setting and cardiopulmonary exercise testing, to see what happens in the lungs of this group of patients when they reach peak exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of sarcoidosis
* Sarcoidosis clinician diagnoses airways involvement
* Aged 18 and above

Exclusion Criteria:

* Current combustible cigarette or electronic cigarette user
* Significant doubt over the diagnosis of sarcoidosis
* Asthma or other airways disease, requiring regular inhaler use
* Contraindication to MRI identified on safety questionnaire
* Recent COVID-19 infection (lateral flow or PCR swab positive within the last 28 days) or ongoing symptoms from COVID-19

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Sarcoidosis patients aged over 18. Non-smokers with no other airways disease or contraindication to MRI.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
Does endobronchial sarcoidosis produce changes, which are appreciable on ventilation MRI and are they temporally stochastic or deterministic. (1) | 12 weeks
  Ventilation defect percentage (VDP) - a measure of amount of the lung which goes unventilated
Does endobronchial sarcoidosis produce changes, which are appreciable on ventilation MRI and are they temporally stochastic or deterministic.(2) | 12 weeks
  Ventilation Coefficient of variation (CV) - a measure of ventilation heterogeneity
Does endobronchial sarcoidosis produce changes, which are appreciable on ventilation MRI and are they temporally stochastic or deterministic. (3) | 12 weeks
  Apparent diffusion coefficient (ADC) and mean linear intercept (LmD) - measurements of the Brownian motion of gas in the acinar airways and surrogate measures of acinar integrity.
Does endobronchial sarcoidosis produce changes, which are appreciable on ventilation MRI and are they temporally stochastic or deterministic. (4) | 12 weeks
  Red blood cell to tissue plasma ratio (RBC:TP) - a measure of the efficiency of gas exchange across the alveoli into the blood.

CONTACTS AND LOCATIONS:
Locations (1):
- University MRI Unit, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No